CLINICAL TRIAL: NCT06740331
Title: Social Cognition, Memory, and Executive Functions in Bipolar Disorder and Major Depressive Disorder
Acronym: COMET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO24114*
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Bipolar Disorder and Major Depressive Disorder
Keywords: Bipolar disorder; major depressive disorder; high-risk individuals; social cognition; executive functions; memory functions
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: participants are assigned to one of two or more groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Bipolar patients (Experimental): Patients with a diagnosis of bipolar disorder
  Interventions: Behavioral: Analysis of social cognition, memory functioning, and executive functioning processes
- Major depressive patients (Experimental): Patients with a diagnosis of major depressive disorder
  Interventions: Behavioral: Analysis of social cognition, memory functioning, and executive functioning processes
- First-degree relatives of bipolar patients (Experimental): First-degree relatives of bipolar patients
  Interventions: Behavioral: Analysis of social cognition, memory functioning, and executive functioning processes
- Bipolar controls (Experimental): Healthy control participants matched to group 1
  Interventions: Behavioral: Analysis of social cognition, memory functioning, and executive functioning processes
- Depressive controls (Experimental): Healthy control participants matched to group 2
  Interventions: Behavioral: Analysis of social cognition, memory functioning, and executive functioning processes
- First-degree controls (Experimental): Healthy control participants matched to group 3
  Interventions: Behavioral: Analysis of social cognition, memory functioning, and executive functioning processes

INTERVENTIONS:
Behavioral: Analysis of social cognition, memory functioning, and executive functioning processes — Investigation of social cognition, memory functioning, and executive processes using a comprehensive clinical and cognitive assessment

SUMMARY:
Bipolar disorder (BD) are common psychiatric disorders often misdiagnosed, leading to delayed treatment. Even during stable phases, individuals with bipolar disorder experience residual cognitive impairments that affect their social functioning and quality of life.

This study aims to explore social cognition deficits (e.g., emotional processing, theory of mind, attribution bias) and their relationship with executive functions (e.g., flexibility, inhibition, working memory) and memory in bipolar disorder and major depressive disorder, ultimately seeking to improve understanding of their functional outcomes.

Social cognition and executive functions in BD are both state- and trait-related. One recent meta-analysis demonstrated impairment in social cognitive domains for manic, depressive, and euthymic bipolar disorders' patients but it remains unclear whether these social cognitive deficits in BD are due to executive functions and/or other confounding effects.

Few studies have investigated the interdependency between these cognitive impairments in these two affective disorders while a better understanding of the link between executive functions and social cognition seems crucial in order to better characterize the nature of patients' deficits and thus their caring.

DETAILED DESCRIPTION:
Bipolar Disorders (BD) and Major Depressive Disorder (MDD) are two of the most common psychiatric disorders worldwide. BD is characterized by severe mood fluctuations (i.e., hypomanic/manic and depressive episodes) and can often be misdiagnosed as MDD, leading to delays in proper diagnosis. This is because the most common initial presentation of BD is a depressive episode. Such delays result in less appropriate care and support.

In addition to delayed diagnoses, the periods between symptomatic episodes, which are considered "stable," are not without challenges. Even during these euthymic periods, individuals often experience residual difficulties that impact their daily functioning. While these periods are viewed as symptom-free, it's clear that individuals still do not experience a significantly improved quality of life. Functional outcomes (e.g., occupational and social functioning) are often impaired and distinguishing between BD and MDD more clearly could improve care and enhance their quality of life. Identifying distinctive markers is essential for improving treatment strategies.

Cognitive functions might serve as trait markers of the disorders because they are impaired both during acute episodes and euthymic phases. These cognitive impairments could also predict functional outcomes in BD. Cognitive profiles may also help distinguish between BD and MDD. While impairments in executive functions, such as the ability to adapt to new situations (e.g., task-switching) and episodic memory (i.e., memory of specific personal events), are present even during euthymic phases of BD, this is not always the case for social cognition (e.g., facial emotion recognition). These cognitive alterations are highly heterogeneous across patients, and identifying their cognitive profiles could provide valuable insights.

Studying the links between cognitive components in BD and MDD may lead to a better understanding how cognitive functions are impacted in these mood disorders, and especially to understand the interactions between these different functions. Additionally, considering clinical symptomatology (e.g., the number of episodes) and other factors (e.g., anxiety, childhood trauma, social support) could offer a more comprehensive understanding of these disorders.

In addition to focusing on these two clinical populations, we will also include first-degree relatives of individuals with bipolar disorder. Indeed, it seems that these relatives may also experience mild cognitive impairments, and we aim to further investigate these hypotheses.

This project aims to better understand social cognition impairments (e.g., emotion processing, theory of mind, attribution bias) and their relationship with verbal episodic memory and executive functions (e.g., working memory, cognitive flexibility) in BD and MDD. It will also explore how these cognitive processes affect functional outcomes in these groups.

A first visit will be dedicated to the collection of clinical data. During the second visit, the investigators will conduct a comprehensive neuropsychological assessment to evaluate executive functions, episodic memory, and all components of social cognition. This protocol will allow the investigators to study all these variables together and to clarify and better understand the connections between them.

ELIGIBILITY:
Inclusion criteria:

* Patients between 18 and 65 years old, men or women
* Having a diagnosis of bipolar disorder or depressive disorder
* No substantial change in treatment for 2 weeks preceding study enrollment
* Being a native French speaker
* Patients enrolled in the national healthcare insurance program
* Consenting to participate to the study

Exclusion criteria:

* The presence of any alcohol use disorder or any other substance use disorder in the last six months, except for tobacco dependence
* A significant general medical illness, including neurological disorders or head trauma
* A sensorial impairment uncorrected (visual and/or hearing)

Group 3: First-degree relatives of bipolar patients

Inclusion criteria:

* Participants between 18 and 65 years old, men or women
* Participants having at least one first-degree relative presenting an bipolar disorder (parents, children, siblings)
* Being a native French speaker
* Patients enrolled in the national healthcare insurance program
* Consenting to participate to the study

Exclusion criteria:

* A diagnosis of schizophrenia or of bipolar disorder or of depressive disorder according to DSM-5 criteria
* The presence of any alcohol use disorder or any other substance use disorder in the last six months, except for tobacco dependence
* A significant general medical illness, including neurological disorders or head trauma
* A sensorial impairment uncorrected (visual and/or hearing)

Group 4, 5, 6: Healthy control participants

Inclusion criteria:

* Participants between 18 and 65 years old, men or women
* Being a native French speaker
* Patients enrolled in the national healthcare insurance program
* Consenting to participate to the study

Exclusion criteria:

* A diagnosis of schizophrenia or of bipolar disorder or of major depressive disorder according to DSM-5 criteria
* The presence of any alcohol use disorder or any other substance use disorder in the last six months, except for tobacco dependence
* Participants having one first-degree relative presenting an bipolar disorder or depressive disorder or schizophrenia according to DSM-5 criteria
* A significant general medical illness, including neurological disorders or head trauma
* A sensorial impairment uncorrected (visual and/or hearing)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2028-01-07 (Estimated); Study Completion 2028-02-07 (Estimated)

PRIMARY OUTCOMES:
Social cognition: facial emotion recognition | Day 0
  Evaluated through Penn Emotion Recognition Task (Emotion Recognition, ER-40). The ER-40 asks participants to assign an emotion to 40 photographs depicting expressions of one of 5 emotions (happiness, sadness, anger, fear and neutral), 4 each of low and high intensity. Are measured the number of correct responses and type of errors.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided